CLINICAL TRIAL: NCT07034066
Title: Study of Hypersensitivity to Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) in Pediatric Population
Brief Title: Pediatric Non-Steroidal Anti-Inflammatory Drugs (NSAID) Allergy Study
Acronym: NSAID-AS
Status: Completed | Type: Observational
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Hospital Sant Joan de Deu (Other)
Responsible Party: Sponsor
Other Study IDs: Sant Joan de Deu Foundation
Record Dates: First submitted 2025-05-29; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-05

CONDITIONS: NSAID; Biomarkers; Phenotyping; Children
Keywords: NSAID-hipersensitivity in children; children drug allergy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 11 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective Cohort: Includes new patients referred to the Pediatric Allergy outpatient clinic with suspected NSAID hypersensitivity.
  Inclusion Criteria:
  Children aged 0-17 years Clinical suspicion of NSAID hypersensitivity
  Exclusion Criteria:
  Refusal to provide informed consent
  At the first outpatient visit:
  A complete medical history and physical exam will be performed The need for DPT (oral/nasal) will be explained to the family Informed consent will be obtained On admission for oral DPT: blood and urine samples will be collected DPT will be conducted via oral route unless the original reaction occurred after intravenous administration Positive DPTs will be followed by sample collection and symptom management A follow-up phone call will be made within 6 months to assess home tolerance
  For patients undergoing nasal DPT, the test will be conducted in the hospital's ENT unit, and follow-up will depend on the result.
- Retrospective Cohort: Includes all patients who underwent a DPT for NSAID hypersensitivity between 2014 and 2021 in the Pediatric Allergy Unit.
  Inclusion Criteria:
  Children aged 0-17 years Completed DPT with the suspected and/or alternative NSAID
  Exclusion Criteria:
  Patients who did not undergo or complete the DPT
  Upon protocol approval, data on all hospital admissions related to NSAID hypersensitivity evaluation (2014-2021) will be requested. Clinical records will be reviewed after pseudonymization, which will be performed by an independent individual, Ms. Silvia del Valle, who will also safeguard the pseudonymization key. This complies with legal requirements for accessing medical records without consent, under CEIm approval, including:
  Functional and technical separation between investigators and data processors Explicit confidentiality and non-reidentification commitment

SUMMARY:
Non-steroidal anti-inflammatory drugs (NSAIDs) are some of the most commonly used medications to treat pain and inflammation. Many are available over the counter and are frequently used in children to reduce fever and relieve pain. Hypersensitivity (HS) to NSAIDs affects an estimated 0.6% to 5.7% of the general population. These reactions can be caused by immune or non-immune mechanisms. In most cases, they fall into two categories: reactions to a single NSAID or to several different NSAIDs.

Currently, the main way to diagnose NSAID hypersensitivity is through a drug provocation test (DPT)-this involves giving the patient the suspected drug under medical supervision to check for a reaction. It's considered the most reliable method. However, diagnosing these reactions in children can be challenging. Symptoms can vary widely, and there are few accurate alternative tests available to replace the DPT.

This study looks for easier ways-like symptoms or lab tests-to diagnose NSAID reactions, so fewer patients need to go through multiple DPT.

DETAILED DESCRIPTION:
Hypersensitivity reactions (HSR) to NSAID in children, although similar to those in adults, present unique challenges in terms of diagnosis and management. While international classification systems are useful, real-world clinical scenarios often fall outside established criteria. Examples include:

* Multiple NSAID HSR involving both cutaneous and respiratory symptoms.
* NSAID-induced anaphylaxis dependent on food intake.
* Immediate selective reactions to more than one NSAID. These scenarios are frequently observed in pediatric patients, highlighting the need for a regional study to evaluate and properly address them.

This is a single-center, ambispective observational study.

Primary Objective:

To describe the clinical characteristics of children with NSAID hypersensitivity.

Secondary Objectives:

1. To describe the different clinical phenotypes and assess age-related differences.
2. To assess tolerance to alternative NSAIDs in patients with confirmed hypersensitivity.
3. To evaluate the usefulness of in vivo and in vitro tests in the diagnostic process.
4. To disseminate study findings.

The study design is based on 2 components:

* Retrospective Component: include participants diagnosed with NSAID HSR, who underwent DPT in the Pediatric Allergy Department at Hospital Sant Joan de Déu between January 2014 and December 2021. Data will be pseudonymized. A waiver of informed consent will be requested due to the long study period, the absence of risk, and the fact that many patients are no longer under follow-up.
* Prospective Component: participants with suspected NSAID HSR were included. Participants will be assessed during outpatient visits, where the following steps will occur:
* In vivo testing, where appropriate, using validated prick and intradermal techniques for paracetamol and metamizole. Controls will include saline (negative) and histamine (positive).
* A DPT will be performed with the suspected medication and/or suitable alternatives, in accordance with standard clinical practice.
* Nasal DPT using a rhinomanometer for patients suspected of NSAID-exacerbated respiratory disease (NERD).
* Families will be informed about the procedures, and informed consent will be obtained.

On the day of the DPT, a blood test (including total IgE, IgG, IgA, IgM, tryptase, IL-6) and urine sample (uLTE4 levels) will be collected.

If the DPT is positive, a second round of blood and urine samples will be collected.

The NSAID to be used in testing are commonly prescribed in pediatric practice and grouped by chemical structure:

Salicylic acid derivatives: Aspirin Para-aminophenol derivatives: Paracetamol (acetaminophen) Propionic acid derivatives: Ibuprofen, naproxen Acetic acid derivatives: Diclofenac Enolic acid derivatives: Pyrazolones, oxicams Fenamates (fenamic acid derivatives) COX-2 inhibitors: Celecoxib

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-17 years
* Completed DPT with the suspected and/or alternative NSAID

Exclusion Criteria:

* Patients who did not undergo or complete the DPT

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of pediatric patients (aged 0 to 17 years) with a clinical suspicion or confirmed diagnosis of hypersensitivity NSAID.
  Retrospective Cohort: Includes all patients who underwent at least one drug provocation test (DPT) for suspected NSAID hypersensitivity between January 2014 and December 2021 at the Pediatric Allergy Department of Hospital Sant Joan de Déu.
  Prospective Cohort: Includes newly referred patients to the outpatient Pediatric Allergy Clinic from August 2022 to December 2024, presenting with clinical symptoms suggestive of NSAID hypersensitivity. Eligibility is determined based on:
  * Clinical manifestations (cutaneous and/or respiratory) following NSAID intake.
  * A high likelihood of an adverse drug reaction based on history.
  * Informed consent signed by parents or legal guardians.
  * Patients with incomplete DPTs or those whose guardians decline consent (for the prospective arm) are excluded.
Sampling Method: Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Clinical characteristics of pediatric patients with NSAID hypersensitivity, based on historical data and development of a diagnostic protocol. | Retrospective arm: review of the medical records took about 4-6 months Prospective arm: from enrollment to DPT, 6-8 months.
  In both the retrospective and prospective arm, the investigators reviewed the medical records of patients who completed DPT. Participant demographic data were reviewed, including age, sex, personal and family history of atopy, and the results of DPTs performed on suspected medications and alternatives if necessary.
  Final phenotypes after DPT were:
  * Cross-intolerance (CI)
  * Selective hypersensitivity (SH)

SECONDARY OUTCOMES:
Differences in clinical features across different pediatric age groups. | Retrospective arm: review of the medical records took about 4-6 months Prospective arm: from enrollment to DPT, 6-8 months.
  In both the retrospective and prospective groups, factors that may predispose to having a confirmed HS based on the clinical history will be analyzed: sex, age, history of atopy, angioedema, rash/urticaria, reason for which the drug is prescribed, having presented more than 1 reaction with the same drug or different NSAIDs.
Rate of tolerance to alternative NSAIDs among patients with confirmed hypersensitivity. | Retrospective arm: review of the medical records took about 4-6 months Prospective arm: from enrollment to DPT, 6-8 months.
  In the retrospective arm, in participants with cross-intolerance, all tolerated high-dose paracetamol and COX-2 inhibitors (meloxicam). Those with selective NSAID HS were tested for tolerance to alternatives from other groups as appropriate.
  In the prospective arm, the investigators do not yet have results.
Diagnostic performance of in vivo and in vitro tests. | Prospective arm: from enrollment to DPT, 6-8 months.
  Both in vivo and in vitro testing were performed in the prospective arm, and DPT is still pending, so the investigators are waiting to complete this in order to analyze the results.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be available beginning 6 months after publication and will remain accessible for 5 years. The results will be available in clinicaltrials.gov with supporting information (Clinical Study Report (CSR)).
Supporting Information: CSR
Time Frame: Data will be available beginning 6 months after publication and will remain accessible for 5 years.
Access Criteria: Data will be shared with qualified researchers affiliated with academic or healthcare institutions, for purposes of academic research or meta-analysis, and can be used for further analysis of the intervention's efficacy, safety profiling, or inclusion in systematic reviews. Study protocol, statistical analysis plan, and informed consent forms (in anonymized format) will also be made available. Requests should be submitted to the corresponding author by email. A data access agreement must be signed, and the research proposal will be reviewed by the study steering committee before approval is granted.
URL: https://www.sjdrecerca.org/es/fundacion/

REFERENCES:
- [Result] Klaewsongkram J, Buranapraditkun S, Mongkolpathumrat P, Palapinyo S, Chantaphakul H. Clinical Characteristics, Urinary Leukotriene E4 Levels, and Aspirin Desensitization Results in Patients With NSAID-Induced Blended Reactions. Allergy Asthma Immunol Res. 2021 Mar;13(2):229-244. doi: 10.4168/aair.2021.13.2.229. PMID 33474858
- [Result] Dona I, Saenz de Santa Maria R, Moreno EM, Bartra J, Torres MJ. An algorithm for the diagnosis and treatment of nonsteroidal antiinflammatory drugs hypersensitivity, 2024 update. Allergy. 2025 Apr;80(4):1183-1186. doi: 10.1111/all.16349. Epub 2024 Oct 4. No abstract available. PMID 39365158
- [Result] Blanca-Lopez N, Haroun-Diaz E, Ruano FJ, Perez-Alzate D, Somoza ML, Vazquez de la Torre Gaspar M, Rivas-Ruiz F, Garcia-Martin E, Blanca M, Canto G. Acetyl Salicylic Acid Challenge in Children with Hypersensitivity Reactions to Nonsteroidal Anti-Inflammatory Drugs Differentiates Between Cross-Intolerant and Selective Responders. J Allergy Clin Immunol Pract. 2018 Jul-Aug;6(4):1226-1235. doi: 10.1016/j.jaip.2017.08.029. Epub 2017 Oct 3. PMID 28986120
- [Result] Cavkaytar O, Arga M. NSAID Hypersensitivity in the Pediatric Population: Classification and Diagnostic Strategies. J Asthma Allergy. 2022 Sep 28;15:1383-1399. doi: 10.2147/JAA.S267005. eCollection 2022. PMID 36199560
- [Result] Kidon M, Blanca-Lopez N, Gomes E, Terreehorst I, Tanno L, Ponvert C, Chin CW, Caubet JC, Soyer O, Mori F, Blanca M, Atanaskovic-Markovic M. EAACI/ENDA Position Paper: Diagnosis and management of hypersensitivity reactions to non-steroidal anti-inflammatory drugs (NSAIDs) in children and adolescents. Pediatr Allergy Immunol. 2018 Aug;29(5):469-480. doi: 10.1111/pai.12915. Epub 2018 Jun 13. PMID 29693290

DOCUMENTS (2):
  • Study Protocol: last version (2024-07-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT07034066/Prot_000.pdf
  • Study Protocol: first version (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT07034066/Prot_001.pdf